CLINICAL TRIAL: NCT05181371
Title: Ultrasound Guided, Continuous Erector Spinae Plane (ESP) Block in Minimally Invasive Thoracic Surgery: Comparing Programmed Intermittent Bolus (PIB) vs Continuous Infusion on Quality of Recovery and Postoperative Respiratory Function
Brief Title: ESP Block in VATS: Programmed Intermittent Bolus Versus Continuous Infusion on Quality of Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mater Misericordiae University Hospital (Other)
Responsible Party: Principal Investigator, Aneurin Moorthy, Anaesthesia Specialist Registrar, Mater Misericordiae University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESP2
Record Dates: First submitted 2021-12-19; First posted 2022-01-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pain, Acute; Surgery
Keywords: Regional Anesthesia; Erector Spinae Block; VATS; Quality of Recovery; Acute pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided ESP Block with Programmed Intermittent Bolus (PIB) (Active Comparator): After induction of general anaesthesia, an ESP catheter will be inserted at the level of T5. A bolus dose of 20 ml 0.25% Levobupicaine will be administered into the ESP space. Two hours post bolus administration, patients will receive programmed intermittent bolus of local anaesthetic: 20mls 0.125% levobupivacaine every two hours.
  Interventions: Procedure: Ultrasound Guided ESP Block with Programmed Intermittent Bolus (PIB) for VATS
- Ultrasound Guided ESP Block with Continuous Infusion (CI) (Active Comparator): After induction of general anaesthesia, an ESP catheter will be inserted at the level of T5. A bolus dose of 20 ml 0.25% Levobupicaine will be administered into the ESP space. Two hours post bolus administration, patients will receive a continuous infusion local anaesthetic: 0.125% levobupivacaine at an infusion rate of 10 ml/hr.
  Interventions: Procedure: Ultrasound Guided ESP Block with Continuous Infusion (CI) for VATS

INTERVENTIONS:
Procedure: Ultrasound Guided ESP Block with Programmed Intermittent Bolus (PIB) for VATS — Programmed Intermittent Bolus (PIB) of Levobupivacaine
  Arms: Ultrasound Guided ESP Block with Programmed Intermittent Bolus (PIB)
Procedure: Ultrasound Guided ESP Block with Continuous Infusion (CI) for VATS — Continuous Infusion (CI) of Levobupivacaine
  Arms: Ultrasound Guided ESP Block with Continuous Infusion (CI)

SUMMARY:
Fascial plane blocks, such as ESP, rely on the spread of local anaesthetic on an interfacial plane, automated boluses may be particularly useful for this group of blocks. However, until recently, ambulatory pumps capable of providing automated boluses in addition to patient-controlled boluses were not widely available. To best of our knowledge, there are no randomised controlled trials comparing continuous infusion versus intermittent bolus strategies for Erector Spinae Plane Block for MITS in terms of patient centred outcomes such as quality of recovery.

DETAILED DESCRIPTION:
Minimally invasive thoracic surgery (MITS) has been shown to reduce postoperative pain, reduce tissue trauma and contribute to better recovery as compared to open thoracotomy. However, it still causes significant acute post-operative pain. Our Mater research group has shown that fascial plane blocks such as the Erector Spinae Plane block (ESP) contribute to post-operative analgesia after MITS. Case reports have described the improved quality of analgesia following ESP using programmed intermittent boluses (PIB) instead of continuous infusion. It is hypothesised that larger, repeated bolus doses provide superior analgesia, possibly as a result of improved spread of the local anaesthetic. Evidence for improved spread of local anaesthetic may be found in one study which demonstrated that PIB increased the number of affected dermatomal levels compared to continuous infusions for continuous paravertebral blocks. Similarly, with regard to labour epidural analgesia, PIB provides better analgesia compared with continuous infusion.

Because fascial plane blocks, such as ESP, rely on the spread of local anaesthetic on an interfacial plane, automated boluses may be particularly useful for this group of blocks. However, until recently, ambulatory pumps capable of providing automated boluses in addition to patient-controlled boluses were not widely available. To the best of our knowledge, there are no randomised controlled trials comparing continuous infusion versus intermittent bolus strategies for Erector Spinae Plane Block for MITS in terms of patient-centered outcomes such as quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female aged > 18
* Able to provide written informed consent
* ASA grade I - V
* VATS surgery
* Weight > 55kg

Exclusion Criteria:

* Absence of or inability to give informed consent
* Pre-existing infection at block site
* Severe coagulopathy
* Allergy to local anaesthesia (or another contraindication to block performance)
* Previous history of opiate abuse
* Pre-existing chronic pain condition
* Pre-existing dementia (due to need to co-operate in completing QoR-15 score day after surgery
* Postoperative admission to ICU for continued ventilation
* BMI > 40 kg/m2

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery (QoR-15) | 24 hours
  Patient centred metric to measure the quality of recovery after surgery. Scale is between 0-150, where '0' refers to poor quality of recovery and '150' refers to excellent quality of recovery

SECONDARY OUTCOMES:
Maximal inspiratory volume | 48 hours
  This will be measured with a calibrated incentive spirometer at the bedside
Area Under the Curve for Verbal Rating Score for pain at rest | 48 hours
  Pain scores (0-10). '0' refers to no pain and '10' refers to severe pain.
Area Under the Curve for Verbal Rating Score for pain on deep inspiration | 48 hours
  Pain scores (0-10). '0' refers to no pain and '10' refers to severe pain.
Time to first intravenous opioid | 48 hours
  Will be measured from immediate postoperative in minutes
Time to first mobilisation | 48 hours
  Will be measured from immediate postoperative in hours
Duration of time in PACU . | 24 hours
  Will be measured from immediate postoperative in minutes
Length of hospital stay | 30 days
  Will be measured from immediate postoperative in days
Quality of Recovery (QoR-15) | 48 hours
  Patient centred metric to measure the quality of recovery after surgery. Scale is between 0-150, where '0' refers to poor quality of recovery and '150' refers to excellent quality of recovery

CONTACTS AND LOCATIONS:
Overall Officials: Donal Buggy, Principal Investigator — Mater University Hospital
Locations (2):
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - St Jame's University Hospital, Dublin

IPD SHARING:
Plan to Share IPD: Yes
Individual Patient Data sharing will be supported with qualified external researchers and supporting clinical documents from eligible studies. All data provided will be coded and anonymised to respect the privacy of patients who have participated in the trial.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5 years
Access Criteria: Publications, reports or query requests from future investigators.

REFERENCES:
- [Background] Finnerty D, Ni Eochagain A, Ahmed M, Poynton A, Butler JS, Buggy DJ. A randomised trial of bilateral erector spinae plane block vs. no block for thoracolumbar decompressive spinal surgery. Anaesthesia. 2021 Nov;76(11):1499-1503. doi: 10.1111/anae.15488. Epub 2021 Apr 20. PMID 33878196
- [Background] Finnerty DT, McMahon A, McNamara JR, Hartigan SD, Griffin M, Buggy DJ. Comparing erector spinae plane block with serratus anterior plane block for minimally invasive thoracic surgery: a randomised clinical trial. Br J Anaesth. 2020 Nov;125(5):802-810. doi: 10.1016/j.bja.2020.06.020. Epub 2020 Jul 11. PMID 32660716
- [Background] Onuoha OC. Epidural Analgesia for Labor: Continuous Infusion Versus Programmed Intermittent Bolus. Anesthesiol Clin. 2017 Mar;35(1):1-14. doi: 10.1016/j.anclin.2016.09.003. Epub 2016 Dec 12. PMID 28131113
- [Background] Ilfeld BM, Gabriel RA. Basal infusion versus intermittent boluses for perineural catheters: should we take the 'continuous' out of 'continuous peripheral nerve blocks'? Reg Anesth Pain Med. 2019 Mar;44(3):285-286. doi: 10.1136/rapm-2018-100262. Epub 2019 Jan 13. No abstract available. PMID 30636717
- [Derived] Eochagain AN, Moorthy A, O'Gara A, Buggy DJ. Ultrasound-guided, continuous erector spinae plane (ESP) block in minimally invasive thoracic surgery-comparing programmed intermittent bolus (PIB) vs continuous infusion on quality of recovery and postoperative respiratory function: a double-blinded randomised controlled trial. Trials. 2022 Sep 21;23(1):792. doi: 10.1186/s13063-022-06726-7. PMID 36131308
- See also: ESP vs PVB — https://doi.org/10.21203/rs.3.rs-703831/v1